CLINICAL TRIAL: NCT04531995
Title: Development of an Artificial Intelligence-based Incident Prediction Algorithm to Improve Cancer Patient Care and Patient Safety
Brief Title: One Million Cancer Treatment Months
Acronym: OMCAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cankado GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: CAN-20-01
Record Dates: First submitted 2020-08-21; First posted 2020-08-31 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Cancer
Keywords: Artificial Intelligence
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CANKADO PRO-React Onco — CANKADO PRO-React Onco is approved as class I medical device within the European Union (registration number DE /CA59 /371/2020-R/Hd) and is compliant with the FDA classification for Mobile Medical Devices (2015) Appendix B. The purpose of CANKADO PRO-React Onco is to be an automated digital support for patients to help them decide how urgent it is to contact the attending physician based on the symptoms they independently record in the system. It supports patients with cancer under systemic, anti-tumor or anti-hormonal therapy in adjuvant, neoadjuvant, post-neoadjuvant or palliative situations. It is unsuitable for patients undergoing radiotherapy, cell and gene therapy, surgical procedures or alternative healing methods.

SUMMARY:
The OMCAT Register aims to provide learning databases in cancer comprising both PRO data using PRO-React and "ground truth" (outcome data verified by the physician during patient examinations). Intelligent learning and knowledge engineering procedures will utilize this PRO data to provide high-quality event prediction algorithms. The ground-truth data enables so-called "supervised learning" techniques of artificial intelligence, because predicted events can be verified with a high level of certainty from ground-truth data.

DETAILED DESCRIPTION:
The next generation of PRO-React by CANKADO is designed to predict impending incident threats at an earlier stage than previously feasible and -- by more timely intervention -- help physicians to eliminate or mitigate the severity of an unfavourable event, reduce the required intensity of countermeasures, or otherwise reduce patient risks.

A highly reliable identification of situations classified as "low-risk" by CANKADO could also enable a more focused utilization of resources as well as enhanced patient comfort and decreased stress, e.g., due to less frequent monitoring visits or reduced need for invasive diagnostics.

The OMCAT Register aims to provide learning databases in cancer comprising both PRO data using PRO-React and "ground truth" (outcome data verified by the physician during patient examinations). Intelligent learning and knowledge engineering procedures will utilize this PRO data to provide high-quality event prediction algorithms. The ground-truth data enables so-called "supervised learning" techniques of artificial intelligence, because predicted events can be verified with a high level of certainty from ground-truth data.

The PRO data of a patient provide what is known in engineering, physics, and statistics as "time series" of observations. The unique feature of PRO time series for applications in cancer is the very high "sampling frequency" (e.g., daily or better) compared to examinations, which generally occur at fixed, and much less frequent intervals. Prediction algorithms based on PRO data would thus be ideally suited to reduce the delay in detecting events, for example, by triggering physician appointments or indicating the need for more intensive medical diagnostics.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 years
* Diagnosed with cancer
* Prescribed CANKADO PRO-React Onco

Exclusion Criteria:

* Lack of consent to study participation or lack of patient's ability to consent
* Enrolled in this trial within a further treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer Patients under systemic, anti-tumor or anti-hormonal therapy in adjuvant, neoadjuvant, post-neoadjuvant or palliative situations with prescribed CANKADO PRO-React Onco will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 166000 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Health Status | 6 months
  Using the EuroQol-visual analogue scale, abbreviated as EQ-VAS Scale, containing values between 100 (best imaginable health) and 0 (worst imaginable health), (answered by patients)
Complaints/Symptoms | 6 months
  Assessed using a question set aligned with the PRO-CTCAE and CTCAE (answered by patients)
Presence or Absence of SAEs | 6 months
  yes/no (answered by physician)
Presence or Absence of dosis reductions | 6 months
  yes/no (answered by physician)
Presence or Absence of treatment interruptions | 6 months
  yes/no (answered by physician)
Presence or Absence of disease progression | 6 months
  yes/no (answered by physician)
Presence or Absence of disease regression | 6 months
  yes/no (answered by physician)
Presence or Absence of death | 6 months
  yes/no (answered by physician)

SECONDARY OUTCOMES:
Cancer type | 6 months
  according to ICD classification
Patient Typology | 6 months
  According to Bloem et al (PMID: 32771005)
Timepoints of patient documentation | 6 months
  The timepoints at which a patient uses the CANKADO System to document patient-reported outcomes are retrieved from the system including date and time
Frequency of patient documentation | 6 months
  The frequency at which a patient uses the CANKADO System to document patient-reported outcomes are calculated using the timepoints of patient documentation

CONTACTS AND LOCATIONS:
Overall Officials: Timo Schinköthe, PhD, Study Director — Cankado GmbH
Locations (4):
- Germany (4):
  - Onkologische Praxis Moers, Moers
  - Ev. Krankenhaus Bethesda Praxis für gynäkologische Onkologie, Mönchengladbach
  - Schwerpunktpraxis für Hämatologie und Onkologie, Soest
  - Hämatologisch-Onkologische Schwerpunktpraxis - Novum medicum, Würzburg